CLINICAL TRIAL: NCT00335556
Title: Treatment of High Risk Renal Tumors: A Groupwide Phase II Study
Brief Title: Combination Chemotherapy, Radiation Therapy, and/or Surgery in Treating Patients With High-Risk Kidney Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AREN0321; NCI-2009-00414 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); COG-AREN0321 (Other: Children's Oncology Group); CDR0000472893 (Other: ClinicalTrials.gov); AREN0321 (Other: Children's Oncology Group); AREN0321 (Other: CTEP); U10CA098543 (NIH)
Record Dates: First submitted 2006-06-08; First posted 2006-06-12 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2017-07-21 (Actual); Status verified 2016-04

CONDITIONS: Childhood Renal Cell Carcinoma; Clear Cell Renal Cell Carcinoma; Clear Cell Sarcoma of the Kidney; Papillary Renal Cell Carcinoma; Rhabdoid Tumor of the Kidney; Stage I Renal Cell Cancer; Stage I Renal Wilms Tumor; Stage II Renal Cell Cancer; Stage II Renal Wilms Tumor; Stage III Renal Cell Cancer; Stage III Renal Wilms Tumor; Stage IV Renal Cell Cancer; Stage IV Renal Wilms Tumor
MeSH Terms: conditions — Carcinoma, Renal Cell; Wilms Tumor | interventions — Doxorubicin; Irinotecan; Surgical Procedures, Operative; Congresses as Topic; Cyclophosphamide; Etoposide; Carboplatin; Dactinomycin; Vincristine; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Surgery (Experimental): Patients with completely resectable stage I-IV RCC undergo surgical resection. Patients with incompletely resectable stage III-IV RCC undergo treatment as per physician's choice.
  Interventions: Procedure: Conventional Surgery
- Treatment (UH-1) (Experimental): Patients receive combination chemotherapy comprising vincristine, doxorubicin hydrochloride, cyclophosphamide, etoposide, and carboplatin. Patients whose primary tumors were initially resected undergo radiotherapy once daily 5 days a week for 4-5½ weeks beginning on day 1 in week 1. Patients with delayed primary tumor resection undergo radiotherapy beginning on day 1 in week 13. If the primary tumor was not previously resected, patients undergo resection, if feasible, in week 13. Patients with unresectable clear cell sarcoma of the kidney (CCSK) receive no further study therapy.
  Interventions: Drug: Doxorubicin Hydrochloride; Procedure: Conventional Surgery; Drug: Cyclophosphamide; Drug: Etoposide; Drug: Carboplatin; Drug: Vincristine Sulfate; Radiation: Radiation Therapy; Other: Laboratory Biomarker Analysis
- Treatment (window/UH-1) (Experimental): Patients receive vincristine IV on days 1 and 8 and irinotecan hydrochloride IV over 30 minutes on days 1-5 and 8-12 (course 1). Patients with progressive disease (PD) are treated with regimen UH-1. Patients with stable disease (SD), partial response (PR), or complete response (CR) receive another course of irinotecan hydrochloride/vincristine window therapy beginning on day 22. After the second course, patients with SD or PD are treated with regimen UH-1 and patients with PR or CR are treated with regimen UH-2.
  Interventions: Drug: Doxorubicin Hydrochloride; Drug: Irinotecan Hydrochloride; Procedure: Conventional Surgery; Drug: Cyclophosphamide; Drug: Etoposide; Drug: Carboplatin; Drug: Vincristine Sulfate; Radiation: Radiation Therapy; Other: Laboratory Biomarker Analysis
- Treatment (UH-2) (Experimental): Patients receive combination chemotherapy comprising vincristine, doxorubicin hydrochloride, cyclophosphamide, etoposide, carboplatin, and irinotecan hydrochloride. Patients whose primary tumors were initially resected undergo radiotherapy as in regimen UH-1 beginning on day 1 in week 1. Patients with delayed primary tumor resection undergo radiotherapy as in regimen UH-1 beginning on day 1 in week 7. If the primary tumor was not previously resected, patients undergo resection, if feasible, in week 7.
  Interventions: Drug: Doxorubicin Hydrochloride; Drug: Irinotecan Hydrochloride; Procedure: Conventional Surgery; Drug: Etoposide; Drug: Carboplatin; Drug: Vincristine Sulfate; Radiation: Radiation Therapy; Other: Laboratory Biomarker Analysis
- Treatment (regimen I) (Experimental): Patients receive vincristine, doxorubicin hydrochloride, cyclophosphamide, and etoposide. Patients whose primary tumors were initially resected (except those with stage I CCSK) undergo radiotherapy as in regimen UH-1 beginning on day 1 in week 1. Patients with delayed primary tumor resection undergo radiotherapy as in regimen UH-1 beginning on day 1 in week 13. If the primary tumor was not previously resected, patients undergo resection, if feasible, in week 13.
  Interventions: Drug: Doxorubicin Hydrochloride; Procedure: Conventional Surgery; Drug: Cyclophosphamide; Drug: Etoposide; Drug: Vincristine Sulfate; Radiation: Radiation Therapy; Other: Laboratory Biomarker Analysis
- Treatment (regimen DD-4A) (Experimental): Patients receive dactinomycin, vincristine, and doxorubicin hydrochloride. Patients whose primary tumors were initially resected undergo radiotherapy as in regimen UH-1 beginning on day 1 in week 1. Patients with delayed primary tumor resection undergo radiotherapy as in regimen UH-1 beginning on day 1 in week 13. If the primary tumor was not previously resected, patients undergo resection, if feasible, in week 13.
  Interventions: Drug: Doxorubicin Hydrochloride; Procedure: Conventional Surgery; Biological: Dactinomycin; Drug: Vincristine Sulfate; Radiation: Radiation Therapy; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Doxorubicin Hydrochloride — Given IV
  Arms: Treatment (UH-1); Treatment (UH-2); Treatment (regimen DD-4A); Treatment (regimen I); Treatment (window/UH-1)
Drug: Irinotecan Hydrochloride — Given IV
  Arms: Treatment (UH-2); Treatment (window/UH-1)
Procedure: Conventional Surgery — Patients undergo resection
  Other Names: surgery, conventional
Drug: Cyclophosphamide — Given IV
  Arms: Treatment (UH-1); Treatment (regimen I); Treatment (window/UH-1)
Drug: Etoposide — Given IV
  Other Names: Lastet
  Arms: Treatment (UH-1); Treatment (UH-2); Treatment (regimen I); Treatment (window/UH-1)
Drug: Carboplatin — Given IV
  Arms: Treatment (UH-1); Treatment (UH-2); Treatment (window/UH-1)
Biological: Dactinomycin — Given IV
  Other Names: Lyovac Cosmegen
  Arms: Treatment (regimen DD-4A)
Drug: Vincristine Sulfate — Given IV
  Other Names: Kyocristine; Oncovin; VCR; Vincasar
  Arms: Treatment (UH-1); Treatment (UH-2); Treatment (regimen DD-4A); Treatment (regimen I); Treatment (window/UH-1)
Radiation: Radiation Therapy — Undergo radiotherapy
  Other Names: Cancer Radiotherapy; Irradiate; Irradiated; Irradiation; RT
  Arms: Treatment (UH-1); Treatment (UH-2); Treatment (regimen DD-4A); Treatment (regimen I); Treatment (window/UH-1)
Other: Laboratory Biomarker Analysis — Correlative studies
  Arms: Treatment (UH-1); Treatment (UH-2); Treatment (regimen DD-4A); Treatment (regimen I); Treatment (window/UH-1)

SUMMARY:
This phase II trial is studying how well combination chemotherapy, radiation therapy, and/or surgery work in treating patients with high-risk kidney tumors. Drugs used in chemotherapy work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving combination chemotherapy together with radiation therapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate whether a treatment regimen containing cyclophosphamide, carboplatin, and etoposide alternating with vincristine, doxorubicin hydrochloride, and cyclophosphamide (regimen UH-1) improves the event-free and overall survival of patients with diffuse anaplastic Wilms' tumor (DAWT) as compared to historical controls.

II. Evaluate, in a phase II "window" study, the antitumor activity of a combination of vincristine and protracted-schedule irinotecan hydrochloride in patients with metastatic DAWT.

III. Evaluate whether regimen UH-1 improves the event-free and overall survival of patients with malignant rhabdoid tumor (MRT) as compared to historical controls.

IV. Maintain the excellent event-free survival of patients with stage I clear cell sarcoma of the kidney (CCSK) without the use of abdominal irradiation.

SECONDARY OBJECTIVES:

I. Describe the outcomes of patients with stage I DAWT or stages I-III focal anaplastic Wilms' tumor (FAWT) treated with vincristine, dactinomycin, doxorubicin hydrochloride, and flank radiation.

II. Describe the outcomes of patients with stage IV FAWT or stage IV CCSK treated with regimen UH-1.

III. Describe event-free and overall survival of children and adolescents with localized renal cell carcinoma (RCC) (including patients with local lymph node involvement) treated with surgical resection without adjuvant therapy.

IV. Describe response rate, event-free survival, and overall survival of patients with unresectable or distantly metastatic RCC treated according to institutional preference.

V. Correlate histologic and molecular cytogenetic findings with outcome in pediatric RCC.

VI. Evaluate the frequency of germline and inherited INI1 mutations in renal and extrarenal MRT and correlate the presence of detectable INI1 mutation with clinical outcome.

VII. Determine the frequency of TP53 mutations in anaplastic Wilms' tumor and correlate the presence of detectable TP53 mutation with clinical outcome.

OUTLINE: This is a multicenter study. Patients are assigned to 1 of 6 treatment regimens according to tumor histology, stage of disease, and response to treatment.

SURGERY (renal cell carcinoma [RCC]): Patients with completely resectable stage I-IV RCC undergo surgical resection. Patients with incompletely resectable stage III-IV RCC undergo treatment as per physician's choice.

REGIMEN UH-1 (stage II-III or stage IV [with no measurable disease] diffuse anaplastic Wilms' tumor [DAWT], stage I-IV malignant rhabdoid tumor [MRT], stage IV focal anaplastic Wilms' tumor [FAWT], or stage IV clear cell sarcoma of the kidney [CCSK]): Patients receive vincristine IV on day 1 in weeks 1-3, 10-12, 13-15, 22-24, and 28-30; doxorubicin hydrochloride IV over 15 minutes on day 1 and cyclophosphamide (CPM2) IV over 15-30 minutes on day 1 in weeks 1, 10, 13, 22, and 28; and cyclophosphamide (at lower doses [CPM1]) IV over 1 hour and etoposide IV over 1 hour on days 1-4 and carboplatin IV over 1 hour on day 1 in weeks 4, 7, 16, 19, and 25. Patients whose primary tumors were initially resected undergo radiotherapy once daily 5 days a week for 4-5½ weeks beginning on day 1 in week 1. Patients with delayed primary tumor resection undergo radiotherapy beginning on day 1 in week 13. If the primary tumor was not previously resected, patients undergo resection, if feasible, in week 13. Patients with unresectable CCSK receive no further study therapy.

IRINOTECAN/VINCRISTINE WINDOW THERAPY* (stage IV DAWT with measurable disease at diagnosis): Patients receive vincristine IV on day 1 and irinotecan hydrochloride IV over 30 minutes on days 1-5 in weeks 1 and 2. Patients with progressive disease (PD) are treated with regimen UH-1. Patients with stable disease (SD), partial response (PR), or complete response (CR) receive another course of irinotecan hydrochloride/vincristine window therapy beginning on day 22. After the second course, patients with SD or PD are treated with regimen UH-1 and patients with PR or CR are treated with regimen UH-2.

NOTE: *Patients who are eligible for but who are unwilling to receive window therapy, receive therapy on regimen UH-1.

REGIMEN UH-2 (DAWT with CR/PR to irinotecan hydrochloride/vincristine window therapy): Patients receive vincristine on day 1 in weeks 1-3, 10, 11, 16-21, 25, 26, 28-30, and 34-36 and doxorubicin hydrochloride and CPM2 as in regimen UH-1 in weeks 1, 16, 19, 28, and 34. Patients also receive CPM1, etoposide, and carboplatin as in regimen UH-1 in weeks 4, 7, 13, 22, and 31 and irinotecan hydrochloride IV over 30 minutes on days 1-5 in weeks 10, 11, 25, and 26. Patients whose primary tumors were initially resected undergo radiotherapy as in regimen UH-1 beginning on day 1 in week 1. Patients with delayed primary tumor resection undergo radiotherapy as in regimen UH-1 beginning on day 1 in week 7. If the primary tumor was not previously resected, patients undergo resection, if feasible, in week 7.

REGIMEN I (stage I-III CCSK): Patients receive vincristine IV on day 1 in weeks 1-3, 5-9, 8-9, 11-14, 19, and 25; doxorubicin hydrochloride IV over 15 minutes on day 1 and cyclophosphamide IV over 1 hour on days 1-3 in weeks 1, 7, 13, 19, and 25; and cyclophosphamide IV and etoposide IV on days 1-5 in weeks 4, 10, 16, and 22. Patients whose primary tumors were initially resected (except those with stage I CCSK) undergo radiotherapy as in regimen UH-1 beginning on day 1 in week 1. Patients with delayed primary tumor resection undergo radiotherapy as in regimen UH-1 beginning on day 1 in week 13. If the primary tumor was not previously resected, patients undergo resection, if feasible, in week 13.

REGIMEN DD-4A (stage I DAWT or stages I-III FAWT): Patients receive dactinomycin IV over 1-5 minutes on day 1 in weeks 1, 7, 13, 19, and 25; vincristine IV on day 1 in weeks 1-10, 13, 16, 19, 22, and 25; and doxorubicin hydrochloride IV over 15 minutes on day 1 in weeks 4,10, 16, and 22. Patients whose primary tumors were initially resected undergo radiotherapy as in regimen UH-1 beginning on day 1 in week 1. Patients with delayed primary tumor resection undergo radiotherapy as in regimen UH-1 beginning on day 1 in week 13. If the primary tumor was not previously resected, patients undergo resection, if feasible, in week 13. Treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically for at least 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed disease of 1 of the following histologic types:

  * Focal anaplastic Wilms' tumor
  * Diffuse anaplastic Wilms' tumor
  * Clear cell sarcoma of the kidney
  * Malignant rhabdoid tumor (renal or extrarenal)
  * Renal cell carcinoma

    * Clear cell
    * Papillary
    * Renal medullary
    * Oncocytoid
    * Sarcomatoid
    * Chromophobe
    * Translocation
    * Collecting duct
    * Carcinoma associated with neuroblastoma
    * Renal cell carcinoma unclassified
* Specimens/materials must be submitted for central review by Day 7
* Patients must begin protocol therapy on AREN0321 by Day 14 after surgery or biopsy (surgery/biopsy is Day 0), unless medically contraindicated
* Karnofsky performance status (PS) must be >= 50 for patients > 16 years if age and Lansky PS must be >= 50 for patients =< 16 years of age
* Patients must not have received systemic chemotherapy or radiation therapy prior to treatment on this study UNLESS they were enrolled on the AREN0532 or AREN0533 studies and received prenephrectomy chemotherapy for what was originally presumed to be favorable histology Wilms tumor; additionally, patients with pediatric RCC who previously received chemotherapy for another type of malignancy (not the RCC) or non-malignant condition may enroll on the study
* Total bilirubin =< 1.5 times upper limit of normal (ULN) for age
* Serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST] or serum glutamic pyruvate transaminase (SGPT) (alanine aminotransferase [ ALT]) < 2.5 times ULN for age
* Shortening fraction of >= 27% by echocardiogram OR ejection fraction of >= 50% by radionuclide angiogram
* Female patients of childbearing age must have a negative pregnancy test
* Female patients who are lactating must agree to stop breast-feeding
* Sexually active patients of childbearing potential must agree to use effective contraception
* All patients and/or their parents or legal guardians must sign a written informed consent
* All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met

Max Age: 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 291 (Actual)
Dates: Start 2006-06; Primary Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Dome, MD, Principal Investigator — Children's Oncology Group
Locations (187):
- United States (161):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of South Alabama, Mobile, Alabama
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - University of Arizona Health Sciences Center, Tucson, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Southern California Permanente Medical Group, Downey, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Miller Children's Hospital, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital Central California, Madera, California
  - Children's Hospital and Research Center at Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Childrens Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - University of California San Francisco Medical Center-Parnassus, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Lombardi Comprehensive Cancer Center at Georgetown University, Washington D.C., District of Columbia
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - Memorial Healthcare System - Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville South, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Miami Children's Hospital, Miami, Florida
  - Baptist Hospital of Miami, Miami, Florida
  - Florida Hospital Orlando, Orlando, Florida
  - UF Cancer Center at Orlando Health, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - Saint Joseph Children's Hospital of Tampa, Tampa, Florida
  - Saint Mary's Hospital, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - Memorial University Medical Center, Savannah, Georgia
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Saint Luke's Mountain States Tumor Institute, Boise, Idaho
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Advocate Children's Hospital-Oak Lawn, Oak Lawn, Illinois
  - Advocate Lutheran General Hospital., Park Ridge, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Southern Illinois University, Springfield, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Saint Vincent Hospital and Health Services, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Kosair Children's Hospital, Louisville, Kentucky
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Maine Children's Cancer Program, Scarborough, Maine
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Michigan State University Clinical Center, East Lansing, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Helen DeVos Children's Hospital at Spectrum Health, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Kalamazoo Center for Medical Studies, Kalamazoo, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - The Childrens Mercy Hospital, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Saint John's Mercy Medical Center, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Nevada Cancer Research Foundation CCOP, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Memorial Hospital, Morristown, New Jersey
  - UMDNJ - Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - University of New Mexico, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - New York University Langone Medical Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Weill Medical College of Cornell University, New York, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Mission Hospital-Memorial Campus, Asheville, North Carolina
  - University of North Carolina, Chapel Hill, North Carolina
  - Carolinas Medical Center, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - The Toledo Hospital/Toledo Children's Hospital, Toledo, Ohio
  - Mercy Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Natalie Warren Bryant Cancer Center at Saint Francis, Tulsa, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center, Portland, Oregon
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Hershey Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Saint Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Palmetto Health Richland, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Greenville Cancer Treatment Center, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - T C Thompson Children's Hospital, Chattanooga, Tennessee
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Texas Tech University Health Science Center-Amarillo, Amarillo, Texas
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine, Houston, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Vermont College of Medicine, Burlington, Vermont
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Childrens Hospital-King's Daughters, Norfolk, Virginia
  - Naval Medical Center - Portsmouth, Portsmouth, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Carilion Clinic Children's Hospital, Roanoke, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - West Virginia University Charleston, Charleston, West Virginia
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin
- Australia (8):
  - John Hunter Children's Hospital, Hunter Regional Mail Centre, New South Wales
  - Sydney Children's Hospital, Randwick, New South Wales
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Royal Children's Hospital-Brisbane, Herston, Queensland
  - Women's and Children's Hospital-Adelaide, North Adelaide, South Australia
  - Royal Children's Hospital, Parkville, Victoria
  - Princess Margaret Hospital for Children, Perth, Western Australia
- Canada (16):
  - Alberta Children's Hospital, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Janeway Child Health Centre, St. John's, Newfoundland and Labrador
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Chedoke-McMaster Hospitals, Hamilton, Ontario
  - Cancer Centre of Southeastern Ontario at Kingston General Hospital, Kingston, Ontario
  - Children's Hospital, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec, Ste-Foy, Quebec
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
- Starship Children's Hospital, Grafton, Auckland, New Zealand
- San Jorge Children's Hospital, San Juan, Puerto Rico

REFERENCES:
- [Derived] Benedetti DJ, Renfro LA, Tfirn I, Daw NC, Kalapurakal JA, Ehrlich PF, Khanna G, Perlman E, Warwick A, Gow KW, Paulino AC, Seibel NL, Grundy P, Fernandez CV, Geller JI, Mullen EA, Dome JS. Treatment and outcomes of clear cell sarcoma of the kidney: A report from the Children's Oncology Group studies AREN0321 and AREN03B2. Cancer. 2024 Jul 1;130(13):2361-2371. doi: 10.1002/cncr.35266. Epub 2024 Feb 23. PMID 38396300

RESULTS

PARTICIPANT FLOW:
Groups:
- Surgery: Surgery Only
- UH-1: Cyclophosphamide/carboplatin/etoposide; vincristine/doxorubicin/cyclophosphomide; x 30 weeks; XRT.
- Window/UH-1: Window therapy of vincristine/irinotecan;Cyclophosphamide/carboplatin/etoposide; vincristine/doxorubicin/cyclophosphomide; x 30 weeks; XRT.
- UH-2: Window therapy of vincristine/irinotecan;Cyclophosphamide/carboplatin/etoposide; vincristine/doxorubicin/cyclophosphomide; x 36 weeks; XRT.
- Regimen I: Vincristine/doxorubicin/cyclophosphamide; cyclophosphamide/etoposide x25 weeks; XRT.
- Regimen DD-4A: Vincristine/dactinomycin/doxorubicin x25 weeks; XRT.
Period: Overall Study
Arm/Group | Surgery | UH-1 | Window/UH-1 | UH-2 | Regimen I | Regimen DD-4A
Started | 68 | 98 | 7 | 10 | 78 | 30
Completed | 66 | 64 | 2 | 5 | 77 | 29
Not Completed | 2 | 34 | 5 | 5 | 1 | 1
Not completed — Death | 0 | 5 | 0 | 0 | 1 | 0
Not completed — Lack of Efficacy | 0 | 19 | 3 | 3 | 0 | 1
Not completed — Physician Decision | 0 | 6 | 2 | 1 | 0 | 0
Not completed — Ineligible | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Refusal of further protocol therapy | 0 | 4 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Surgery | UH-1 | Window/UH-1 | UH-2 | Regimen I | Regimen DD-4A | Total
Number analyzed (Participants) | 68 | 98 | 7 | 10 | 78 | 30 | 291
Age, Continuous [Mean (Standard Deviation); unit: Months] | 148.53 (51.74) | 52.39 (40.09) | 68.95 (97.64) | 54.04 (19.71) | 34.10 (31.10) | 54.29 (32.72) | 70.60 (60.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 55 | 5 | 7 | 31 | 11 | 137
  Male | 40 | 43 | 2 | 3 | 47 | 19 | 154
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 8 | 0 | 2 | 15 | 4 | 34
  Not Hispanic or Latino | 63 | 88 | 6 | 8 | 63 | 25 | 253
  Unknown or Not Reported | 0 | 2 | 1 | 0 | 0 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 0 | 0 | 3 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Black or African American | 22 | 17 | 1 | 2 | 13 | 5 | 60
  White | 40 | 72 | 5 | 8 | 55 | 22 | 202
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 4 | 8 | 1 | 0 | 7 | 3 | 23

OUTCOME MEASURES:

1. Primary Outcome: Event-Free Survival of Patients With Diffuse Anaplastic Wilms' Tumor (DAWT)
Description: Compare the outcome of patients treated with alternating CyCE/VDCy chemotherapy (with or without vincristine/irinotecan cycles) to a fixed outcome based on that seen for similar patients treated with NWTS-5 (NCT00002610).
Time Frame: 4 years
Population: Eligible patients with Stage II-IV DAWT.
Measure: Number (95% Confidence Interval); unit: Percentage of 4-year OS
Arm/Group | UH-1 | Window/UH-1 | UH-2
Number analyzed (Participants) | 52 | 4 | 10
Percentage of 4-year OS | 76.1 [62.5 to 89.6] | 25.0 [0 to 67.4] | 87.5 [64.6 to 100.0]
Statistical Analysis 1: Comparison: UH-1 vs Window/UH-1 vs UH-2; The event-free survival distributions of patients with Stage II-IV diffuse anaplastic Wilms' tumor on AREN0321 and NWTS-5 (NCT00002610) were compared using the log-rank test; Test type: Other; p = .0199, Log Rank; Log Rank Test Statistic = 5.4190

2. Primary Outcome: Long-term Survival of Patients With Stage I-IV Malignant Rhabdoid Tumors
Description: The outcome of these patients will be compared with a fixed outcome based on that seen for similar patients treated with NWTS-5 regimen (NCT00002610).
Time Frame: 4 years
Population: Eligible patients with Stage I-IV rhabdoid tumor.
Measure: Number (95% Confidence Interval); unit: Percentage of 4-year OS
Groups:
- UH-1: Cyclophosphamide/carboplatin/etoposide; vincristine/doxorubicin/cyclophosphamide; x 30 weeks; XRT.
Arm/Group | UH-1
Number analyzed (Participants) | 36
Percentage of 4-year OS | 38.9 [20.1 to 57.7]
Statistical Analysis 1: Comparison: UH-1; The overall survival distributions of patients with Stage I-IV malignant rhabdoid tumors on AREN0321 and National Wilms Tumor Study-5 -- Treatment of Relapsed Patients, A National Wilms Tumor Study Group Phase III Study (NCT00002610) were compared using the log-rank test; Test type: Other; p = .3478, Log Rank; Log Rank Test Statistic = .8814

3. Primary Outcome: Response Rate
Description: Criteria for response assessed by three-dimensional measurement: Complete Response (CR), Disappearance of all index lesions and non-index lesions. No new lesions; Partial Response (PR), At least a 65% decrease in the sum of the volumes of the index lesions. No new lesions; Response rate (RR) = CR+PR of patients who received window therapy.
Time Frame: Up to 2 months
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Combined Window/UH-1 and UH-2: Combine window/UH-1 and UH-2 for response rate monitoring for window therapy.
Arm/Group | Combined Window/UH-1 and UH-2
Number analyzed (Participants) | 17
Percentage of participants | 71 [49 to 92]

4. Primary Outcome: Event Free Survival Probability
Description: Event-free survival will be informally compared to that seem for similar patients treated on NWTS-5 (NCT00002610).
Time Frame: 4 years
Population: Eligible patients with Stage I focal and diffuse anaplastic Wilms tumor.
Measure: Number (95% Confidence Interval); unit: Percent Probability 4 Year EFS
Arm/Group | Regimen DD-4A
Number analyzed (Participants) | 18
Percent Probability 4 Year EFS | 100.0 [100.0 to 100.0]
Statistical Analysis 1: Comparison: Regimen DD-4A; The event-free survival distributions of patients with Stage I focal and diffuse anaplastic Wilms tumors on AREN0321 and National Wilms Tumor Study-5 -- Treatment of Relapsed Patients, A National Wilms Tumor Study Group Phase III Study (NCT00002610) were compared using the log-rank test; Test type: Other; p = .0570, Log Rank; Log Rank Test Statistic = 3.6216

5. Primary Outcome: Toxicity Rate
Description: Percentage of participants with Grade 4 cardiac toxicities, Grade 4 Sinusoidal Obstruction Syndrome (SOS), and treatment-related deaths determined using CTCAE v4.
Time Frame: Up to 4 years
Population: Eligible patients treated after Amendment 3A for arms UH-1, UH-2, and Window/UH-1.
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Groups:
- Combined UH-2, UH-1, Window/UH-1: Combined UH-1, UH-2, and Window/UH-1 for revised-UH toxicity monitoring
Arm/Group | Combined UH-2, UH-1, Window/UH-1
Number analyzed (Participants) | 61
Percentage of patients
  Cardiac toxicities | 4.9 [0 to 10.3]
  Treatment-related deaths | 4.9 [0 to 10.3]
  Sinusoidal Obstruction Syndrome | 0 [0 to 0]

6. Secondary Outcome: Number of Patients With INI1 Mutations in Renal and Extrarenal Malignant Rhabdoid Tumor by Fluorescent in Situ Hybridization
Time Frame: At baseline
Population: Eligible patients with reported INI1 mutation data.
Measure: Number; unit: Count participants
Arm/Group | UH-1 | Window/UH-1
Number analyzed (Participants) | 26 | 1
Count participants | 23 | 1

7. Secondary Outcome: Frequency of TP53 Mutations
Time Frame: At baseline
Population: The analysis was supplanted by an analysis done as part of the TARGET initiative on NWTS-5 sample as a result no TP53 data was collected on AREN0321.
Groups:
- UH-1: Cyclophosphamide/carboplatin/etoposide; vincristine/doxorubicin/cyclophosphomide;x 30 weeks; XRT.
- Window/UH-1: Window therapy of vincristine/irinotecan;Cyclophosphamide/carboplatin/etoposide;vincristine/doxorubicin/cyclophosphomide; x 30 weeks; XRT.
Arm/Group | UH-1 | Window/UH-1 | UH-2 | Regimen DD-4A
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Groups:
- UH-1: Cyclophosphamide/carboplatin/etoposide;vincristine/doxorubicin/cyclophosphomide; x 30 weeks; XRT
- Window/UH-1: Window therapy of vincristine/irinotecan; Cyclophosphamide/carboplatin/etoposide;vincristine/doxorubicin/cyclophosphomide; x 30 weeks; XRT"
- Regimen DD-4A: Vincristine/dactinomycin/doxorubicin x25 weeks; XRT"
Arm/Group | Surgery | UH-1 | Window/UH-1 | UH-2 | Regimen I | Regimen DD-4A
Serious Adverse Events (participants affected / at risk) | 2/66 | 19/98 | 3/7 | 0/10 | 3/78 | 1/30
Other Adverse Events (participants affected / at risk) | 0/66 | 81/98 | 5/7 | 9/10 | 7/78 | 1/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Surgery (N=66) | UH-1 (N=98) | Window/UH-1 (N=7) | UH-2 (N=10) | Regimen I (N=78) | Regimen DD-4A (N=30)
10300-Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
11100-Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
11300-Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
11600-Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
14900-Ascites (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
15000-Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
17400-Blood bilirubin increased (Investigations) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
19200-Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
20000-Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
20100-Cardiac disorders - Other specify (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
24100-Creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
24600-Death NOS (General disorders) | 0 (0) | 5 (5) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
24700-Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
34000-Fibrinogen decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
37200-General disorders and administration site conditions (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
39000-Heart failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
43100-Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
43300-Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
43500-Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
43600-Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
43900-Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
44200-Ileal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
44800-Infections and infestations - Other specify (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
51700-Left ventricular systolic dysfunction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
52600-Lipase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
53100-Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
55700-Multi-organ failure (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
58000-Neoplasms benign malignant and unspecified (incl cy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
58100-Nervous system disorders - Other specify (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
60600-Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
65800-Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
65900-Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
66000-Pleural hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
66300-Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
66400-Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
68700-Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
69000-Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
71500-Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
73700-Sepsis (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
78300-Sudden death NOS (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
81200-Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
87900-Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
88200-Weight gain (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Surgery (N=66) | UH-1 (N=98) | Window/UH-1 (N=7) | UH-2 (N=10) | Regimen I (N=78) | Regimen DD-4A (N=30)
10100-Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
10200-Abdominal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
10300-Abdominal pain (Gastrointestinal disorders) | 0 (0) | 6 (6) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
10700-Acidosis (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
11100-Acute kidney injury (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
11300-Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
11400-Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
11600-Alanine aminotransferase increased (Investigations) | 0 (0) | 9 (10) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
13100-Anaphylaxis (Immune system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
13200-Anemia (Blood and lymphatic system disorders) | 0 (0) | 4 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
13500-Anorexia (Metabolism and nutrition disorders) | 0 (0) | 20 (22) | 2 (3) | 2 (2) | 3 (4) | 0 (0)
14100-Apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
14900-Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
15000-Aspartate aminotransferase increased (Investigations) | 0 (0) | 8 (8) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
15400-Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
17200-Blood and lymphatic system disorders - Other specif (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
17400-Blood bilirubin increased (Investigations) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
20000-Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
20500-Catheter related infection (Infections and infestations) | 0 (0) | 7 (7) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
22100-Colitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
22200-Colonic fistula (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
22300-Colonic hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
24100-Creatinine increased (Investigations) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
24300-Cystitis noninfective (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
24700-Dehydration (Metabolism and nutrition disorders) | 0 (0) | 9 (10) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
25700-Diarrhea (Gastrointestinal disorders) | 0 (0) | 10 (11) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
25800-Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
27600-Dysphagia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
27800-Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
28200-Edema face (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
29400-Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
29500-Enterocolitis infectious (Infections and infestations) | 0 (0) | 4 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
29700-Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
31200-Esophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
32400-Facial nerve disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
33300-Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 56 (86) | 3 (5) | 8 (12) | 4 (6) | 0 (0)
33900-Fever (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
36400-Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
36700-Gastrointestinal disorders - Other specify (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
37500-GGT increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
38900-Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
39100-Hematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
39300-Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
40000-Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
40600-Hepatobiliary disorders - Other specify (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
41200-Hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
41300-Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
41400-Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 4 (5) | 1 (1) | 2 (5) | 0 (0) | 0 (0)
41600-Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
41800-Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
42100-Hypertension (Vascular disorders) | 0 (0) | 8 (9) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
42600-Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 4 (4) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
42700-Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
42900-Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
43100-Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 14 (19) | 3 (4) | 1 (1) | 0 (0) | 0 (0)
43200-Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
43300-Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 8 (8) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
43500-Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 5 (7) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
43600-Hypotension (Vascular disorders) | 0 (0) | 8 (8) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
43900-Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 6 (6) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
44800-Infections and infestations - Other specify (Infections and infestations) | 0 (0) | 44 (77) | 4 (4) | 4 (13) | 1 (3) | 0 (0)
46300-Intra-abdominal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
48400-Investigations - Other specify (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
51700-Left ventricular systolic dysfunction (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
52600-Lipase increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
53100-Lung infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
53500-Lymphedema (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
53700-Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
53900-Malabsorption (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
55600-Mucositis oral (Gastrointestinal disorders) | 0 (0) | 9 (9) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
55700-Multi-organ failure (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
56900-Myocarditis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
57600-Nausea (Gastrointestinal disorders) | 0 (0) | 5 (6) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
58100-Nervous system disorders - Other specify (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
58300-Neutrophil count decreased (Investigations) | 0 (0) | 6 (8) | 0 (0) | 1 (1) | 2 (3) | 0 (0)
59600-Oral hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
59700-Oral pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
60100-Otitis media (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
60600-Pain (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
60700-Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
61800-Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
62500-Pelvic infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
63100-Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
63900-Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
64100-Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
64200-Peritoneal infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
65200-Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
65300-Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
65800-Platelet count decreased (Investigations) | 0 (0) | 5 (7) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
65900-Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
66300-Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
66500-Portal hypertension (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
68300-Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
68700-Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
69000-Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
69200-Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
72700-Right ventricular dysfunction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
73700-Sepsis (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
73900-Serum amylase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
74600-Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
74700-Skin and subcutaneous tissue disorders - Other spec (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
75200-Skin infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
75700-Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
76000-Small intestine infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
76400-Soft tissue infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
79600-Thromboembolic event (Vascular disorders) | 0 (0) | 3 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
81800-Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
81900-Typhlitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
82300-Upper respiratory infection (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
83100-Urinary tract infection (Infections and infestations) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
83600-Urine output decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
86400-Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
87900-Vomiting (Gastrointestinal disorders) | 0 (0) | 9 (9) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
88300-Weight loss (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
88500-White blood cell decreased (Investigations) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
88900-Wound infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior Sponsor approval.